CLINICAL TRIAL: NCT03741465
Title: "The Anatolian Sitting Neuraxial Position Technique"; is it Beneficial? A Prospective Clinical Comparison Trial Via Ultrasonography
Brief Title: A New Neuraxial Position Technique " The Anatolian Sitting Position- Sitting Fetal Cross-legged"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Fatma Ferda Kartufan, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: YeditepeU
Record Dates: First submitted 2018-10-26; First posted 2018-11-15 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Anesthesia, Conduction
Keywords: neuraxial anesthesia positioning technique; Anatolian sitting position; sitting cross-legged position; sitting fetal position; ultrasonography; numerical rating scale

STUDY DESIGN:
Intervention Model Description: Systematic randomization was made from 150 volunteers, and 50 participants were chosen.
  All 50 participants were planned to sit on the stretcher in both of the two positioning techniques sequentially (one after another). The two positioning techniques are 1) sitting fetal position-" the SFP" ( a traditional position ) and 2) sitting fetal cross-legged-" the ASP" ( a new position, named as " Anatolian sitting position"). The investigator was planned to record all of the participants' anatomical measurements in both of those positioning techniques evaluated via ultrasonography. After each position participants were planned to evaluate each positioning technique's comfort by 5-point numerical rating scale from minimum 1 meaning "poor" to maximum 5 meaning "excellent."
Who Masked: Outcomes Assessor
Masking Description: The ultrasonography was made by a consultant radiologist (M.D.) Although the consultant didn't know which position was for control and which was the one the study evaluates. Although investigators were trying to mask the outcomes assessor; the consultant saw the positions because there is no way to hide the sitting positions of the participants. So there is a paradox if the consultant is masked or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The SFP technique (Active Comparator): In the SFP neuraxial positioning technique, fifty participants were planned to sit on the stretcher facing the wall of the sonography room and turned back to the consultant Radiologist with legs hanging freely, forearms on the lap and hand are on the knees. The position is completed with the back curved in the fetal position. Then the USG is performed by the consultant Radiology M.D. in maximum 2 hours time to each participant, and the 5-point NRS evaluation is done by each participant in maximum 30 minutes time until the study ends within 24 weeks.
  Interventions: Procedure: The SFP technique
- The ASP technique (Experimental): In the ASP neuraxial positioning technique, the same fifty participants were planned to sit on the same part of the stretcher facing the wall of the sonography room and turned back to the consultant Radiologist with legs crossed, forearms of the participants are on the lap and hands are on the knees, and the position is completed with the back curved in the fetal position.Then the USG is performed by the consultant Radiology M.D. in maximum 2 hours time to each participant, and the 5-point NRS evaluation is done by each participant in maximum 30 minutes time until the study ends within 24 weeks.
  Interventions: Procedure: The ASP technique

INTERVENTIONS:
Procedure: The SFP technique — The USG, and the 5-point NRS evaluation in the SFP
  Arms: The SFP technique
Procedure: The ASP technique — The USG, and the 5-point NRS evaluation in the ASP
  Arms: The ASP technique

SUMMARY:
A prosperous neuraxial anesthesia positioning ensures a raised chance of successful needle placement. The primary aim is to compare "The Anatolian sitting position-ASP" with "The Sitting Fetal Position-SFP" sonographically. Secondary aim is to compare their comfort.

DETAILED DESCRIPTION:
Fifty participants were included to this prospective, randomized, consecutive controlled clinical study. Six parameters were evaluated in each position; subcutaneous tissue (ST), skin to spinous process (S-SP), transverse diameters of bilateral paraspinal muscles (left paraspinal muscle [LPM] and right paraspinal muscle [RPM]), interspinous gap opening (ISGO), mean of bilateral paraspinal muscles (MPM). The change of every measurement recorded via ultrasonography (USG) according to the positioning techniques (the Anatolian Sitting Position [ASP] could also be named as "sitting fetal cross-legged position" and the Sitting Fetal Position [SFP] which is a traditional sitting position) were also calculated. The calculations are explained briefly in primary outcomes (including the change of ASP-SFP in ST, S-SP, LPM, RPM, MPM, ISGO). Stretcher comfort (SC), position comfort (PC), lumbar comfort (LC), and abdominal comfort (AC) were evaluated by the participants with the 5-point Numerical Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* healty and adult volunteers,
* must be able to do the sitting fetal cross-legged position ( ASP ),
* must be able to do the sitting fetal position ( SFP ).

Exclusion Criteria:

* BMI higher than 40,
* Lumbar hernia,
* Scoliosis,
* History of spine surgery,
* History of trauma,
* History of lower back pain,
* Arthropathy {especially pelvic or knee problems},
* Could not be able to do one or both of the two neuraxial position techniques.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Interspinous gap opening (ISGO) measurement in the ASP | For the ASP technique, ISGO is measured in the first 10 minutes(mins.) time, for each participant, through study completion.
  the wideness measurement of the ISGO in millimeters via ultrasonography (USG) in the ASP
Left paraspinal muscle (LPM) measurements in the ASP | For the ASP technique, LPM is measured in between 10mins. and 20mins. time, for each participant, through study completion.
  the diameter measurement of the LPM in millimeters via ultrasonography in the ASP
Right paraspinal muscle (RPM) measurements in the ASP | For the ASP technique, RPM is measured in between 20mins. and 30mins. time, for each participant, through study completion.
  the diameter measurement of the RPM in millimeters via ultrasonography in the ASP
The mean of bilateral paraspinal muscles (MPM) in the ASP | For the ASP technique, MPM measurement is planned to be done in between 30mins. and 40mins. time, for each participant, through study completion.
  Measured by ( [LPM+RPM]/2) in millimeters in the ASP
Subcutaneous tissue (ST) measurements in the ASP | For the ASP technique, ST measurement is planned to be done in between 40mins. and 50mins. time, for each participant, through study completion.
  the thickness measurement of the subcutaneous tissue in millimeters via ultrasonography in the ASP
The skin to spinous process (S-SP) measurements in the ASP | For the ASP technique, S-SP measurement is planned to be done in between 50mins. and 1 hour(hr.) time, for each participant, through study completion.
  the depth measurement of the skin to spinous process in millimeters via ultrasonography in the ASP
Interspinous gap opening (ISGO) measurement in the SFP | For the SFP technique, ISGO measurement is planned to be done, right after NRS evaluation of the ASP, in between 1hr.10mins. and 1hr.20mins. time, for each participant, through study completion.
  the wideness measurement of the ISGO in millimeters via ultrasonography in the SFP
Left paraspinal muscle (LPM) measurements in the SFP | For the SFP technique, LPM measurement is planned to be done in between 1hr.20mins. and 1hr.30mins. time, for each participant, through study completion.
  the diameter measurement of the LPM in millimeters via ultrasonography in the SFP
Right paraspinal muscle (RPM) measurements in the SFP | For the SFP technique, RPM measurement is planned to be done in between 1hr.30mins. and 1hr.40mins. time, for each participant, through study completion.
  the diameter measurement of the RPM in millimeters via ultrasonography in the SFP
The mean of bilateral paraspinal muscles (MPM) in the SFP | For the SFP technique, MPM measurement is planned to be done in between 1hr.40mins. and 1hr.50mins. time, for each participant, through study completion.
  Measured by ( [LPM+RPM]/2) in millimeters in the SFP
Subcutaneous tissue (ST) measurements in the SFP | For the SFP technique, ST measurement is planned to be done in between 1hr.50mins. and 2hrs. time, for each participant, through study completion.
  the thickness measurement of the subcutaneous tissue in millimeters via ultrasonography in the SFP
The skin to spinous process (S-SP) measurements in the SFP | For the SFP technique, S-SP measurement is planned to be done in between 2hrs. and 2hr.10mins. time, for each participant, through study completion.
  the depth measurement of the skin to spinous process in millimeters via ultrasonography in the SFP
the change of ISGO (ISGO ASP-SFP) | ISGO in the ASP is measured in the first 10mins., and ISGO in the SFP is measured in between 1hr.10 mins. and 1hr.20mins. time, through study completion.
  Measured by calculation; ([ISGO in the ASP in millimeters]-[ISGO in the SFP in millimeters])
the change of LPM (LPM ASP-SFP) | LPM in the ASP is measured in between 10mins. and 20mins. time, and LPM in the SFP is measured in between 1hr.20mins and 1hr.30mins. time, through study completion.
  Measured by calculation; ([LPM in ASP in millimeters]-[LPM in SFP in millimeters])
the change of RPM (RPM ASP-SFP) | RPM in the ASP is measured in between 20mins. and 30mins. time, and RPM in the SFP is measured in between 1hr.30mins. and 1hr.40mins. time, through study completion.
  Measured by calculation ([RPM in ASP in millimeters]-[RPM in SFP in millimeters])
the change of MPM (MPM ASP-SFP) | MPM in the ASP is measured in between 30mins. and 40mins. time, and MPM in the SFP is measured in between 1hr.40mins and 1hr.50mins. time, through study completion.
  Measured by calculation ([MPM in ASP in millimeters]-[MPM in SFP in millimeters])
the change of ST (ST ASP-SFP) | ST in the ASP is measured in between 40mins. and 50mins. time, and in the SFP is measured in between 1hr.50mins and 2hrs. time, through study completion.
  Measured by calculation ([ST in ASP in millimeters]-[ST in SFP in millimeters])
the change of S-SP (S-SP ASP-SFP) | S-SP in the ASP is measured in between 50mins. and 1hr. time, and S-SP in the SFP is measured in between 2 hrs. and 2hrs.10mins. time, through study completion.
  Measured by calculation ([S-SP in ASP in millimeters]-[S-SP in SFP in millimeters])

SECONDARY OUTCOMES:
Comfort evaluation in the ASP via 5-point numerical rating scale (NRS) | NRS measurement is planned to be done right after the ASP position in between 1hr. and 1hr.10mins. time, for each participant, through study completion.
  Comfort evaluation of the ASP technique is planned to be done by the participant right after USG. The 5-point NRS includes 5 scale. The minimum scale is"1" means poor, "2" means fair, "3" means good, "4" means very good, and the maximum scale is "5" means excellent.
Comfort evaluation in the SFP via 5-point numerical rating scale (NRS) | NRS measurement is planned to be done right after the SFP position in between 2hrs.10mins. and 2hrs.20mins. time, for each participant, through study completion.
  Comfort evaluation of the SFP technique is planned to be done by the participant right after USG. The 5-point NRS includes 5 scale. The minimum scale is"1" means poor, "2" means fair, "3" means good, "4" means very good, and the maximum scale is "5" means excellent.

CONTACTS AND LOCATIONS:
Overall Officials: ferda kartufan, Principal Investigator
Locations (1):
- Yeditepe University hospital, Istanbul, İçerenköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dimaculangan DP, Mazer JA, Maracaja-Neto LF. Sonographic evaluation of lumbar interlaminar space opening in a variety of patient body positions for optimal neuraxial anesthesia delivery. J Clin Anesth. 2016 Nov;34:159-65. doi: 10.1016/j.jclinane.2016.03.045. Epub 2016 May 6. PMID 27687365